CLINICAL TRIAL: NCT07220590
Title: Bridging the Gap: Implementing A Powered Mobility Intervention Into Early Childhood Settings for Young Children With Cerebral Palsy (GMFCS IV-V)
Brief Title: Implementing Powered Mobility in Early Childhood Settings for Children With Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Bethany Sloane, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1K23HD119273-01 (NIH)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy Children; Motor Disabilities; Developmental Disability; Rehabilitation; Early Intervention; Assistive Technology
Keywords: Power Mobility; Implementation Science; Community-engaged research; Caregiver coaching; Pediatric Rehabilitation
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Powered Mobility Intervention (Experimental): This mixed-methods feasibility trial includes one experimental arm in which all participants receive the powered mobility intervention following a structured therapist training. Trained physical and occupational therapists participate in one to two days of in-person training to learn how to implement the intervention with children with cerebral palsy (GMFCS IV-V) and their caregivers in early childhood settings. Following training, therapists identify eligible child-caregiver dyads from their caseloads and conduct twelve biweekly home-based intervention sessions over six months. Each session focuses on mobility opportunities, caregiver coaching, and integration of powered mobility into daily routines using the Permobil Explorer Mini device. All sessions are video recorded for fidelity monitoring and qualitative analysis.
  Interventions: Behavioral: Therapist Training on Powered Mobility Implementation; Behavioral: Powered Mobility Intervention for Child-Caregiver Dyads

INTERVENTIONS:
Behavioral: Therapist Training on Powered Mobility Implementation — Therapists participate in a structured, evidence-based training on implementing powered mobility interventions for children with cerebral palsy (GMFCS IV-V) in early childhood settings. Training consists of one to two days of in-person sessions focused on knowledge transfer, therapist confidence, self-efficacy, and use of caregiver coaching and routines-based strategies. The training is co-designed with a community advisory board of administrators, therapists, and caregivers to ensure contextual relevance and feasibility.
Behavioral: Powered Mobility Intervention for Child-Caregiver Dyads — Following therapist training, participating therapists deliver a six-month powered mobility intervention to children with cerebral palsy (GMFCS IV-V) and their caregivers. Therapists conduct twelve biweekly home-based sessions focused on providing mobility opportunities, caregiver coaching, and integration of powered mobility into daily routines. The intervention uses the Permobil Explorer Mini device to facilitate self-initiated mobility. All sessions are audio-video recorded for fidelity monitoring and qualitative analysis.

SUMMARY:
The goal of this clinical trial is to learn if a therapist training program can help providers in Part C Early Childhood Settings use powered mobility (PM) with young children who have cerebral palsy (Gross Motor Function Classification System Levels IV-V). The study will also look at whether this training is practical and useful for therapists, families, and children.

The main questions it aims to answer are:

1. Can therapists successfully use the training to provide powered mobility interventions in home and early childhood settings?
2. Do families and children find the intervention acceptable and helpful?
3. What benefits do children show in mobility, participation, and engagement after using powered mobility?

In this study, therapists and families will:

1. Take part in a training program about how to use powered mobility with young children
2. Use powered mobility devices (Permobil Explorer Mini) with children during everyday routines
3. Complete surveys, interviews, and observations about their experiences

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of physical disability in childhood. Children classified at Gross Motor Function Classification System (GMFCS) Levels IV-V experience significant limitations in mobility and typically require assistive technology to move independently. These early months, between 12-36 months, are a critical period for brain development and learning. Without access to independent mobility, children with CP have fewer opportunities to explore, communicate, and engage socially, which can contribute to secondary developmental delays.

Power mobility (PM) devices, such as the Permobil Explorer Mini, provide opportunities for self-initiated exploration of a child's environment. Research has shown that access to PM in early childhood can promote cognitive, social, and motor development, while also supporting participation in family and community life. Despite this growing evidence base, PM use in Part C Early Childhood Settings is infrequent and inconsistent. Many families never receive the option of PM during their child's first years. Barriers include a lack of provider training, limited availability of devices, uncertainty about service delivery models, and the perception that PM should be delayed until school age.

This study directly addresses these gaps by developing and testing a training program for Early Childhood Setting providers to deliver PM interventions with young children with CP (GMFCS IV-V). The project uses a community-engaged, implementation science approach to ensure that the intervention is not only clinically meaningful but also feasible and sustainable within real-world Part C Early Childhood Setting systems.

The research is guided by three aims:

1. Identify provider needs and barriers through surveys and focus groups with providers.
2. Co-design a training program with input from a Community Advisory Board that includes clinicians, families, administrators and researchers. This process ensures that the training reflects real-world challenges and priorities.
3. Conduct a feasibility trial to test the training program with providers and families of young children with CP.

The feasibility trial will combine implementation and child-level outcomes in an effectiveness-implementation hybrid design. Implementation outcomes will include acceptability, appropriateness, feasibility, and fidelity, using validated measures such as the Acceptability of Intervention Measure (AIM), Feasibility of Intervention Measure (FIM), and Implementation Appropriateness Measure (IAM). Fidelity will be examined through session recordings and coding of adherence to intervention strategies.

The intervention itself consists of therapist training in PM use, assessment, and caregiver coaching. Providers will be introduced to the Explorer Mini and will learn strategies to embed mobility into family routines. Therapists will then coach families to use PM with their children during everyday activities, both in the home and community. The emphasis is on real-world use, giving children opportunities to explore, make choices, and participate in their environments.

Child outcomes will include mobility, engagement, and participation, measured through caregiver report, standardized assessments, and observational coding of video-recorded sessions. Family experiences will be assessed through surveys and semi-structured interviews, to better understand acceptability and perceived benefits of PM.

This study is expected to generate critical pilot data on how PM interventions can be implemented in Part C Early Childhood settings, a setting where they are currently underutilized. By focusing on both therapist training and family engagement, this project bridges the gap between evidence and practice. Findings will inform larger-scale trials and lay the groundwork for integrating PM into standard Early Childhood setting services, ensuring that children with CP and significant motor impairments have earlier opportunities to move, explore, and participate fully in daily life.

ELIGIBILITY:
Inclusion Criteria:

Children:

1. Diagnosis of cerebral palsy or similar motor impairment
2. Gross Motor Function Classification System (GMFCS) Levels IV-V
3. Age 12 to 32 months at enrollment
4. Enrolled in early intervention services

Caregivers:

1. Parent or legal guardian of an enrolled child participant
2. Age 18 years or older
3. English- or Spanish-speaking
4. Able and willing to participate in home-based data collection, including caregiver coaching sessions, completion of surveys, and video-recorded sessions
5. Able to provide informed consent

Therapists:

1. Licensed physical therapist or occupational therapist
2. Employed at participating early intervention or early childhood special education settings
3. Provide services to children with cerebral palsy or motor delays
4. No prior powered mobility intervention training required
5. Willing to complete powered mobility implementation training and participate in study assessments

Exclusion Criteria:

1. Inability or unwillingness to provide informed consent
2. Inability to complete required study procedures

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability, Appropriateness, and Feasibility | Post-intervention (after 6 months of intervention).
  Therapist and caregiver perceptions of the powered mobility intervention's acceptability, appropriateness, and feasibility, measured using three validated implementation outcome measures:
  Acceptability of Intervention Measure (AIM) Intervention Appropriateness Measure (IAM) Feasibility of Intervention Measure (FIM) Each measure consists of 4 items rated on a 5-point Likert scale (1 = completely disagree to 5 = completely agree). Total scores range from 4 to 20 for each measure, with higher scores indicating greater acceptability, appropriateness, or feasibility of the intervention. Mean scores will be calculated for each scale.
Therapist Knowledge Transfer, Confidence, and Self-Efficacy | Pre-training and immediately post-training (within 1 week).
  Change in therapist knowledge, confidence, and self-efficacy related to powered mobility implementation, measured using a study-specific therapist questionnaire administered via REDCap. Items are rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores will be calculated, with higher scores indicating greater knowledge, confidence, and self-efficacy. Change scores will be computed from pre-training to post-training.
Caregiver Feasibility of Device and Strategy Use | Biweekly during 6-month intervention period.
  Caregiver-reported feasibility of using the powered-mobility device and implementing facilitating strategies, assessed biweekly with a brief questionnaire. Frequency and mean feasibility ratings over time.
Therapist Intervention Fidelity | Per intervention session throughout the 6-month intervention period.
  Degree to which therapists deliver the powered mobility intervention as intended, assessed through video-coded observations using a structured fidelity checklist and established coding framework. Fidelity ratings capture adherence, dosage, quality of delivery, participant responsiveness, and program differentiation. Mean percentage of fidelity checklist items completed as intended across sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany M Sloane, PT, DPT, PhD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Northwest Regional Education Service District, Hillsboro, Oregon
  - Multnomah Early Childhood Program, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
This is a small, early-stage feasibility study involving young children with cerebral palsy. Given the sensitive nature of pediatric data and the limited sample size, individual participant data will not be shared outside of the study team. However, de-identified, aggregate findings will be disseminated through peer-reviewed publications, conference presentations, and collaboration with community and clinical partners

REFERENCES:
- [Background] Sabet A, Feldner H, Tucker J, Logan SW, Galloway JC. ON Time Mobility: Advocating for Mobility Equity. Pediatr Phys Ther. 2022 Oct 1;34(4):546-550. doi: 10.1097/PEP.0000000000000939. Epub 2022 Aug 4. PMID 35943383
- [Background] Sloane BM, Kenyon LK, Logan SW, Feldner HA. Caregiver perspectives on powered mobility devices and participation for children with cerebral palsy in Gross Motor Function Classification System level V. Dev Med Child Neurol. 2024 Mar;66(3):333-343. doi: 10.1111/dmcn.15718. Epub 2023 Jul 28. PMID 37515376
- [Background] Feldner HA, Logan SW, Otieno S, Fragomeni A, Kono C, Riordan K, Sloane B, Kenyon LK. Short-Term Powered Mobility Intervention Is Associated With Improvements in Development and Participation for Young Children With Cerebral Palsy: A Randomized Clinical Trial. Phys Ther. 2025 Jan 8;105(1):pzae152. doi: 10.1093/ptj/pzae152. PMID 39450982
- [Background] Kenyon LK, Jones M, Livingstone R, Breaux B, Tsotsoros J, Williams KM. Power mobility for children: a survey study of American and Canadian therapists' perspectives and practices. Dev Med Child Neurol. 2018 Oct;60(10):1018-1025. doi: 10.1111/dmcn.13960. Epub 2018 Jun 28. PMID 29956320
- [Background] Kenyon LK, Hostnik L, McElroy R, Peterson C, Farris JP. Power Mobility Training Methods for Children: A Systematic Review. Pediatr Phys Ther. 2018 Jan;30(1):2-8. doi: 10.1097/PEP.0000000000000458. PMID 29252826